CLINICAL TRIAL: NCT01815203
Title: Does Caffeine Consumption Improve Response Inhibition to Food Cues?
Brief Title: Caffein Consumption and Response Inhibition
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uppsala University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: PH2013a
Record Dates: First submitted 2013-03-18; First posted 2013-03-20 (Estimated); Last update posted 2013-09-25 (Estimated); Status verified 2013-09

CONDITIONS: Eating Behavior; Obesity
Keywords: Caffeine effects; Inhibitory control
MeSH Terms: conditions — Feeding Behavior; Obesity | interventions — Caffeine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Caffeine (Experimental): Administration of one gelatin capsule containing 200-300 mg of caffeine with subsequent cognitive tasks and food test.
  Interventions: Drug: Caffeine
- Placebo (Placebo Comparator): Administration of placebo (one gelatin capsule containing starch) with subsequent cognitive tasks and food test.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Caffeine — Administration of one gelatin capsule containing 200-300 mg of caffeine with subsequent cognitive tasks and food test.
  Arms: Caffeine
Drug: Placebo — Administration of placebo with subsequent cognitive tasks and food test.
  Arms: Placebo

SUMMARY:
With the abundance of energy-dense foods that are designed for ease of consumption in the current environment, it is of importance to better understand the factors that may undermine the control of energy intake at healthy levels.

One of the factors that is potentially important in response inhibition is caffeine.

The aim is to assess the direct effects of caffeine on response inhibition, using a No Go/Go-task. We will also assess whether the presentation of food cues, i.e. as words or as pictures, modulate response inhibition different in restrained vs. non-restrained eaters.

DETAILED DESCRIPTION:
In a blinded, randomized cross-over design, participants will receive either a capsule with caffeine or placebo at two separate occasions whereupon study tasks will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Only males
* 18 ≤ 35 years
* Healthy (self rated)
* Used to drink caffeine
* Used to eat breakfast regularly (≥ 5 times a week).
* Non-smokers

Exclusion Criteria:

* BMI outside the range of 18,5 ≤ 25
* hypersensitivity for the ingredients of the foods under study
* being a vegan or vegetarian. Participants reported not using products that are artificially sweetened, nor sugar in coffee and/or tea
* Presence of any chronically disease and/or treatment with medication

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2013-03; Primary Completion 2013-07 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Inhibition control | 20 min
  Measurement inhibition control via a computer test (NoGo-Go task.

SECONDARY OUTCOMES:
Food test | 20 min
  Measure of participants food intake.

OTHER OUTCOMES:
Blood sample | 5 min (1 sample)
  Blood glucose assessment in order to confirm fasted condition prior to study experiments.

CONTACTS AND LOCATIONS:
Overall Officials: Pleunie Hogenkamp, PhD, Principal Investigator — Uppsala University
Locations (1):
- Uppsala University, Uppsala, Sweden